CLINICAL TRIAL: NCT06165094
Title: Effect of Cervical Paraesophageal Lymph Node Metastasis Versus Supraclavicular Lymph Node Metastasis on the Overall Survival of Patients With Thoracic Esophageal Squamous Cell Carcinoma: An Observational Study
Acronym: ECPLNMvsSLNM
Status: Completed | Type: Observational
Sponsor: Sichuan Cancer Hospital and Research Institute (Other)
Responsible Party: Principal Investigator, Yongtao Han, MD, Sichuan Cancer Hospital and Research Institute
Other Study IDs: SCCH-TS2206; 2023YFQ0056 (Other Grant/Funding Number: Sichuan Key Research and Development Project from Science and Technology Department of Sichuan Province)
Record Dates: First submitted 2023-12-03; First posted 2023-12-11 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Esophageal Cancer
Keywords: oesophageal squamous cell carcinoma; cervical paraesophageal lymph node metastasis; supraclavicular lymph node metastasis; lymphadenectomy; esophagectomy
MeSH Terms: conditions — Esophageal Neoplasms; Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Diagnosed with supraclavicular LNM: There was no intervention(s) in any group
- Diagnosed with paraesophageal LNM: There was no intervention(s) in any group

SUMMARY:
The goal of this observational study is to learn about in health conditions of ESCC. The main question[s] it aims to answer are:

•Lymph node metastasis(LNM) in cervical paraesophageal or supraclavicular which influence OS more.

Participants will describe the main status quo after surgery

Researchers will compare Lymph node metastasis(LNM) in cervical paraesophageal and supraclavicular to see if dead.

DETAILED DESCRIPTION:
Demographic and pathologic data, including gender, age, pathological T stage, pathological N stage, 8th tumor-node-metastasis (TNM) stage, tumor location, tumor grade, lymphovascular invasion, perineural invasion, LNM, cervical paraesophageal LNM, supraclavicular LNM, and radical resection, were collected from the Sichuan Cancer Hospital and Institute Esophageal Cancer Case Management (SCH-ECCM) database.

ELIGIBILITY:
The inclusion criteria were as follows:

* patients who had undergone esophagectomy and
* patients who exhibited LNM in the supraclavicular region.

The exclusion criteria:

* tumor location outside the thoracic region,
* pathological examination results confirming the presence of non-squamous cell carcinoma, - patients with both cervical paraesophageal LNM and supraclavicular LNM, or
* those with missing required data

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Demographic and pathologic data, including gender, age, pathological T stage, pathological N stage, 8th tumor-node-metastasis (TNM) stage, tumor location, tumor grade, lymphovascular invasion, perineural invasion, LNM, cervical paraesophageal LNM, supraclavicular LNM, and radical resection, were collected from the Sichuan Cancer Hospital and Institute Esophageal Cancer Case Management (SCH-ECCM) database.
Sampling Method: Non-Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2009-01-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Overall survival | 2009.01.01-2017.12.30
  OS was calculated from the month and year of surgery until the time of death or the last follow-up in March 2021.

CONTACTS AND LOCATIONS:
Locations (1):
- Sichaun cancer hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No